CLINICAL TRIAL: NCT07003477
Title: Biomarkers Based EArly Diagnosis of STroke Subtype Cohort, Bio-EAST
Brief Title: Biomarkers Based EArly Diagnosis of STroke Subtype Cohort（Bio-EAST）
Acronym: Bio-EAST
Status: Recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai Sixth People's Hospital, Affiliated to Shanghai Jiao Tong University (Unknown); Shanghai 7th People's Hospital (Other); Huashan Hospital (Other); Shanghai Zhongshan Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: Bio-EAST
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: stroke; Intracerebral hemorrhage; GFAP (glial fibrillary acidic protein); Pre-hospital diagnosis
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human peripheral blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intracranial hemorrhage, ICH: Patients diagnosed with hemorrhagic stroke by clinical gold standard. Detect the peripheral blood biomarkers，and the results were compared with the clinical gold standard.
  Interventions: Diagnostic Test: Detection of peripheral blood biomarkers
- Non-hemorrhagic stroke: Patients diagnosed with non-hemorrhagic stroke by clinical gold standard. Detect the peripheral blood biomarkers，and the results were compared with the clinical gold standard.
  Interventions: Diagnostic Test: Detection of peripheral blood biomarkers

INTERVENTIONS:
Diagnostic Test: Detection of peripheral blood biomarkers — Peripheral blood samples were collected from patients suffering from acute stroke. The concentration of the biomarker glial fibrillary acidic protein (GFAP) was then detected. This was aimed at differentiating between hemorrhagic stroke and non - hemorrhagic stroke. Time - concentration curves were constructed, thereby offering a novel potential approach for the rapid identification of stroke types within ambulances.

SUMMARY:
Intracerebral hemorrhage carries high rates of mortality and disability, imposes a significant societal burden. Based on findings from our previous multicenter randomized controlled clinical trial (INTERACT4), we revealed that initiating intensive blood pressure reduction therapy within 2 hours of onset in ambulances can markedly enhance the prognosis of patients with intracerebral hemorrhage. Nevertheless, the lack of rapid pre-hospital diagnostic technology hinders its clinical application and promotion. Given that glial fibrillary acidic protein (GFAP), as a biomarker, has been clinically validated for its high specificity in diagnosing intracerebral hemorrhage, this project aims to leverage an industry-academia-research collaborative development model in partnership with Shanghai Jinguan Technology Co., Ltd. By focusing on the urgent need for rapid diagnosis in stroke emergency care, this project will integrate clinical resources from hospitals with technological advantages in product development from the industry. Through resource sharing and complementary strengths, we aim to develop GFAP rapid detection technology with single-molecule sensitivity utilizing internationally advanced silicon photonics technology. Our objectives further include establishing a Chinese cohort to validate the reliability of GFAP in diagnosing intracerebral hemorrhage and conducting multicenter randomized controlled clinical trials to ascertain the efficacy and safety of GFAP-guided pre-hospital intensive blood pressure reduction for patients with intracerebral hemorrhage. This study also aimed to explore other biomarkers to be combined with GFAP in order to improve its sensitivity in detecting ICH.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Suspected stroke at emergency department arrival (FAST score ≥ 2 points, must include limb weakness);
3. Time of stroke symptom onset/last known normal within 3 hours.

Exclusion Criteria:

1. Coma - no response to tactile or verbal stimuli;
2. Severe comorbidities (such as tumors, severe COPD, severe heart failure, requiring assistance with daily living [unable to walk independently]);
3. History of epilepsy or onset with seizure;
4. Recent history of head trauma (< 7 days);
5. Blood glucose < 2.8 mmol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project plans to collect 2 cases per week from each participating medical center (such as Shanghai East Hospital, Zhongshan Hospital, and Huashan Hospital). We anticipate enrolling at least 527 patients. Blood samples will be collected from each patient at 2 time points, resulting in approximately 1,054 specimens in total.
Sampling Method: Non-Probability Sample
Enrollment: 527 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
stroke subtype | Upon arrival at the hospital for the first time
  Cerebral hemorrhage diagnosed by head CT

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided